CLINICAL TRIAL: NCT03342573
Title: Cosentyx (Secukinumab) for the Treatment of Adult Onset Pityriasis Rubra Pilaris: A Single Arm, Open-label Exploratory Trial
Brief Title: Cosentyx (Secukinumab) for the Treatment of Adult Onset Pityriasis Rubra Pilaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jason Sluzevich MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-006987
Record Dates: First submitted 2017-10-18; First posted 2017-11-17 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: PITYRIASIS RUBRA PILARIS
MeSH Terms: conditions — Pityriasis Rubra Pilaris | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Cosentyx (Secukinumab) for the treatment of adult onset pityriasis rubra pilaris
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Patients with a biopsy proven diagnosis of PRP
  Interventions: Drug: Cosentyx

INTERVENTIONS:
Drug: Cosentyx — Cosentyx 300 mg SQ week 0-4, then every q4 weeks for a total of 28 weeks.
  Other Names: Secukinumab

SUMMARY:
The primary objective of this study is to assess the potential effectiveness of Cosentyx in the treatment of adult-onset Pityriasis Rubra Pilaris or PRP.

ELIGIBILITY:
Inclusion Criteria

Informed subject consent will be obtained from those patients meeting the following inclusion criteria:

* Male and female patients 18 years or older.
* Clinical and/or histopathological diagnosis of PRP
* Candidate for systemic therapy (PASI ≥ 10)
* Body surface area of involvement ≥ 10%
* Good general health as confirmed by medical history
* Patients who are willing and capable of cooperating to the extent and degree required by the protocol; and
* Patients who read and sign an approved informed consent for this study

Exclusion Criteria

Patients are to be excluded based on the following criteria:

* Vulnerable study population
* Pregnant or nursing women
* Women planning a pregnancy within the study period
* Human immunodeficiency virus (HIV) positivity
* Known history of adverse reaction to Cosentyx
* Known history of hepatitis B, hepatitis C, or tuberculosis
* Personal or family history of inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
PASI-75 | 28 weeks
  Psoriasis Area and Severity Index (PASI)-75 response rate: the number of study participants with a PASI percent improvement from baseline of ≥ 75%. As no formalized disease severity assessment scoring exists for PRP, the PASI score was selected given the phenotypic overlap between psoriasis and PRP

SECONDARY OUTCOMES:
PASI-90 | 28 weeks
  PASI-90 response rate: the number of study participants with a PASI percent improvement from baseline of ≥ 90%
DLQI | 28 weeks
  Dermatology Quality of Life Index - mean change before and after treatment
PGA | 28 weeks
  Physician Global assessment - mean change before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jason C Sluzevich, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boudreaux BW, Pincelli TP, Bhullar PK, Patel MH, Brumfiel CM, Li X, Heckman MG, Pittelkow MR, Mangold AR, Sluzevich JC. Secukinumab for the treatment of adult-onset pityriasis rubra pilaris: a single-arm clinical trial with transcriptomic analysis. Br J Dermatol. 2022 Nov;187(5):650-658. doi: 10.1111/bjd.21708. Epub 2022 Jul 15. PMID 35701384
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials